CLINICAL TRIAL: NCT04480359
Title: The Clinical Research of the Traditional Chinese Medicine Bawei Shenqi Pill in the Treatment of the Kidney Yang Deficiency Type of Ankylosing Spondylitis
Brief Title: Bawei Shenqi Pill in the Treatment of Ankylosing Spondylitis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, maojianchun, professor, Shanghai University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Bawei Shenqi Pill
Record Dates: First submitted 2020-07-16; First posted 2020-07-21 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-07

CONDITIONS: Ankylosing Spondylitis
Keywords: Bawei Shenqi Pill; ankylosing spondylitis; clinical research
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Meloxicam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bawei Shenqi group (Active Comparator): participants should administrate both Bawei Shenqi Pill and Meloxicam tablets
  Interventions: Drug: Bawei Shenqi Pill; Drug: Meloxicam
- placebo group (Placebo Comparator): participants should administrate both Bawei Shenqi Pill placebo and Meloxicam tablets
  Interventions: Drug: Bawei Shenqi Pill placebo; Drug: Meloxicam

INTERVENTIONS:
Drug: Bawei Shenqi Pill — 5.1g, once a day, 3month, oral
  Other Names: Experimental:Bawei Shenqi group
  Arms: Bawei Shenqi group
Drug: Bawei Shenqi Pill placebo — 5.1g, once a day, 3month, oral
  Other Names: Placebo Comparator: placebo group
  Arms: placebo group
Drug: Meloxicam — 7.5mg, once a day, 3 month, oral
  Other Names: Experimental:Bawei Shenqi group; Placebo Comparator: placebo group

SUMMARY:
The purpose of this study is to determine whether Bawei Shenqi Pill is effective in the treatment of active ankylosing spondylitis (AS).

DETAILED DESCRIPTION:
Ankylosing spondylitis is a chronic inflammatory disease, which mainly invades sacroiliac joint, spinal osteoid process, paraspinal soft tissue and peripheral joints, and can be accompanied by extraarticular manifestations, in severe cases, spinal deformity and ankylosis can occur. The overall prevalence rate of ankylosing spondylitis in China is about 0.3%, the peak of which is 20 to 30 years old. although the prevalence rate is not high, the disability rate is high, and the patients with ankylosing spondylitis are mainly young people of childbearing age, which are in a critical period of work and study. If the disease can not be controlled smoothly, it will seriously affect its learning and work efficiency, image appearance and even the ability of daily life.

Bawei Shenqi Pill originates from Zhang Zhongjing's synopsis of the Golden Chamber, is the representative prescription of warming and tonifying kidney yang, and is also suitable for the pathogenesis of ankylosing spondylitis "deficiency of kidney yang". The purpose of this study was to observe the therapeutic effect of Bawei Shenqi Pill on ankylosing spondylitis of kidney-yang deficiency type through a randomized controlled clinical study. To clarify the effect of Bawei Shenqi Pill on disease activity, joint function, TCM syndrome integral and quality of life in patients with ankylosing spondylitis, and to provide basis for the treatment of ankylosing spondylitis with Bawei Shenqi Pill.

ELIGIBILITY:
Inclusion Criteria:

* Compliance with New York standards revised in 1984
* Syndrome differentiation of traditional Chinese medicine for deficiency of kidney-yang
* 18 to 70 years of age, male and female
* Being able to understand or sign an informed consent form

Exclusion Criteria:

* Other spondyloarthropathy that does not meet the diagnostic criteria of ankylosing spondylitis, and TCM syndrome differentiation does not belong to kidney-yang deficiency type.
* Age is out of range
* Do not agree to participate in this topic or can not participate in the whole process
* Complicated with other rheumatic diseases or other seronegative spondyloarthropathy.
* Pregnant, lactating women and patients with serious visceral diseases, mental disorders and severe extraarticular manifestations, such as heart, lung, liver, kidney or hematopoietic system.
* Have had myocardial infarction or stroke, congestive heart failure and active digestive tract ulcer patients.
* Those who had received other research drugs three months before screening.
* Inability or unwillingness to provide informed consent or failure to comply with test requirements.
* The researchers believe that it is not suitable for the owners of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-08-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
BASDAI | 12weeks
  Bath Ankylosing Spondylitis Disease Activity Index
BASFI | 12weeks
  Bath Ankylosing Spondylitis Functional Index
CRP | 12weeks
  C-reactive protein
ESR | 12weeks
  Erythrocyte sedimentation rate
Range of motion | 12weeks
  occipital wall distance, chest expansion distance, finger ground distance, Schober test

SECONDARY OUTCOMES:
SF-36 | at baseline and at 3 months
  SF- 36 scale for quality of life assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Longhua Hospital Affiliated to Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided